CLINICAL TRIAL: NCT00854698
Title: Long-Term Effects of Aortic Valve Mismatch on Functional Ability and Remodeling the Left Ventricular After Aortic Valve Replacement Mechanics
Brief Title: Long-Term Effects of Aortic Valve Mismatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4199; 2008-A00663-52
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: THE LEFT VENTRICULAR REMODELING AFTER MECHANICAL AORTIC VALVE REPLACEMENT
Keywords: THE LEFT VENTRICULAR REMODELING AFTER MECHANICAL AORTIC VALVE REPLACEMENT; exercise training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group with MVA (Experimental)
  Interventions: Other: exercise training
- group without MVA (Other)
  Interventions: Other: subjects are asked to exercise during 20 or 30 minutes

INTERVENTIONS:
Other: exercise training — subjects are asked to exercise 20 or 30 minutes.
  Arms: Group with MVA
Other: subjects are asked to exercise during 20 or 30 minutes — subjects are asked to exercise during 20 or 30 minutes
  Arms: group without MVA

SUMMARY:
The real impact of the existence of an aortic valve mismatch after aortic valve replacement in various studies conducted so far is a source of controversy. There is currently no long-term impact of the aortic valve mismatch on the reversal of left ventricular remodeling and its impact functional.To evaluate these effects of aortic valve mismatch on abilities to the effort, the quality of life and the regression of left ventricular hypertrophy long term after a aortic valve replacement, conducting a new study is fundamental. This study is even more essential in patients with a young life expectancy theoretical long and physical activity.Our study aims to determine whether the existence of an aortic valve mismatch has an influence on: The functional capacity to the effort by measuring the maximum oxygen consumption during a stress test (VO2 max) The reversal of left ventricular remodeling (cardiac ultrasound doppler), diastolic dysfunction (cardiac ultrasound and Doppler measurement Brain Natriuretic Peptide (BNP). This study will analyse these data in patients who received youth a VAN by mechanical aortic valve prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient major ≤ 60 years at the time of the aortic valve replacement.
* Patient affiliated with a social security
* Consent dated and signed by the investigator and the subject
* Subject having been informed of the results of the visit prior aortic valve replacement by mechanical prosthesis for pure aortic narrowing.
* Fraction left ventricular ejection ≥ 50%, when aortic valve replacement and at the time of inclusion.
* Aortic insufficiency at aortic valve replacement associated <II / IV.
* aortic valve replacement exclusive (no gestures associated: coronary bypass, enlargement of the ring, another valve surgery,…).
* Coronarography normal at the aortic valve replacement.
* Normal renal function.
* No history of heart failure episode in the previous month inclusion.
* No indication against a stress test on bicycle ergometric

Exclusion Criteria:

* Refusal of the patient to be included in the study.
* History of cardiac surgery under extra body movement before and / or after the aortic valve replacement.
* Aortic insufficiency associated with the time of the transaction> II / IV.
* Chronic respiratory insufficiency.
* Track cancer or cancer evolving.
* Evolutionary Osteoarthritis of the lower limbs or widespread.
* Myopathy device.
* Alteration higher making it impossible to carry out the test effort and response to the questionnaire on the quality of life.
* Coronaropathy documented.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
variations in VO2 max during an effort | 1 year

SECONDARY OUTCOMES:
Study the impact of a MVA after RVA by mechanical prosthesis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Petit-Eisenmann Hélène, MD, Principal Investigator — not affiliated
Locations (1):
- CHRU, Nouvel Hôpital Civil, Service de chirurgie cardio-vasculaire, Strasbourg, France

REFERENCES:
- [Result] Petit-Eisenmann H, Epailly E, Velten M, Radojevic J, Eisenmann B, Kremer H, Kindo M. Impact of Prosthesis-Patient Mismatch on Long-term Functional Capacity After Mechanical Aortic Valve Replacement. Can J Cardiol. 2016 Dec;32(12):1493-1499. doi: 10.1016/j.cjca.2016.02.076. Epub 2016 Mar 8. PMID 27297001